CLINICAL TRIAL: NCT02149004
Title: Translational Research Platform of the TTU HIV of the German Center for Infection Research (DZIF)
Brief Title: German Centre for Infection Research HIV Translational Platform
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: German Center for Infection Research (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Dr. med. Jörg Janne Vehreschild, Coordinating Investigator, University Hospital of Cologne
Other Study IDs: DZIF_HIV
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: Human immunodeficiency virus (HIV); Prevention; Long-term life; Cure; Cohort
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquids, tissue, and pathogens from consenting patients will be stored in a decentral biobank.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Site Bonn
- Site Heidelberg
- Site Munich
- Site Hamburg
- Site Hannover
- Site Cologne
- Site Freiburg
- Site Frankfurt
- Site Essen

SUMMARY:
Despite major advances in therapy and management, HIV/AIDS continues to be a major cause of infectious disease morbidity and mortality on a global scale. The discovery of effective antiretroviral treatment has turned HIV infection into a manageable chronic disease in most patients with access to care. However, the different economic and epidemiologic situation in developing and developed countries requires different research priorities, so that three main challanges are universal and in focus of research of the DZIF HIV Translational Platform:

* Prevention of HIV infection
* Long-term life with HIV
* HIV cure

The "Translation Reserach HIV" will bring together clinical researchers in HIV infection in order to develop new treatment options to the above mentioned main challanges. It will take advantage of existing expertise (e.g. basic science, novel targets for treatment and HIV eradiation) of the partner sites. This platform is necessary because Germany's HIV research has suffered in the past from a lack of integration between its excellent basic science and clinical research. In addition, there was too little integration into networks that address the main international challenges. There is an urgent need to link these research strands through dedicated structures emphasising the translation of preclinical results into new therapies.

DETAILED DESCRIPTION:
Structure

The DZIF HIV Translational Platform belongs to the HIV the Thematic Translational Units (TTUs) of the German Centre for Infection Research (DZIF), which is founded by the Federal Ministry of Education and Research (BMBF). The national, multi-centre structure of the DZIF bringing together selceted universities, university hospitals, and non-university research institutes and translational efforts focussing on distinct infectious diesease-related health problems are co-ordinated by the TTUs. The TTU HIV is located in six DZIF partner sites in Germany: Bonn-Cologne, Brunswick-Hannover, Gießen-Marburg-Langen, Hamburg, Heidelberg, Munich.

Mission and Objectives

Prevention of HIV:

The main tools for effective prevention include vaccines, microbicides, preventive therapy and induction of behavioral change. Currently, few groups in Germany have specific preclinical expertise in this area. This expertise needs to be further developed and integrated in the DZIF to be able to implement internationally competitive HIV vaccine and microbicide programmes.

Long-term life with HIV:

This challenge is equally relevant for the developing and developed world. DZIF researchers have made many internationally visible contributions to management of HIV infection in the past. They have extensive experience in clinical studies in the HIV field and have played a major role in the clinical development of new drugs for HIV therapy (e.g. maraviroc, raltegravir). They are also intensively involved in the establishment of clinical guidelines for management of HIV infection.

HIV cure:

Antiretroviral therapy can completely suppress HIV replication below the limit of detection for sustained periods of time, but cannot eradicate the virus from silent reservoirs. Accordingly, life-long therapy is needed and interruption of therapy always leads to resurgence of viral spread and disease. Several approaches have been suggested to eliminate silently infected cells or the HIV genomes integrated in these cells. These approaches are currently mostly at the stage of basic research or early preclinical development and need to be developed in the translational chain. While significant knowledge exists about the nature of silent reservoirs, the number and clonality of viral integration sites is currently largely unknown and needs to be further investigated to develop virus eradication strategies and therapies.

The aim of the DZIF HIV Translational Platform is to comprehensively and collaboratively analyze the above mentioned aspects by using cohorts of HIV infected patients in different stages and with different courses of disease. These cohorts have been established by the participating partner sites, which will be coordinated and extended by the focus site in Bonn-Cologne.

This study protocol is the framework and platform for future substudies.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients HIV positive and who are treated in one of the six partner sites
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-04; Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of new HIV infections in Germany | Up to 20 years
  Overall long-term goal of the platform is to develop a translation strategy for the preclinical results concerning HIV prevention from all German research groups with outstanding expertise. Specific outcome measures will be detailed in future subprojects.

SECONDARY OUTCOMES:
Incidence of chronic organ failure and malignant diseases in HIV infected patients | Up to 20 years
  Overall long-term goal of this platform is to focus on co-infections, organ damage and malignant diseases. Research on identifying new correlates of protection and long term viral control will contribute to improved management of HIV infection. Specific outcome measures will be detailed in future subprojects.

OTHER OUTCOMES:
Sustained viral response rate 12 months after discontinuation of ART | Up to 20 years
  Overall long-term goal of this platform is to eliminate silently infected cells or the HIV genomes integrated in these cells. These approaches are currently mostly at the stage of basic research or early preclinical development and need to be developed in the translational chain. Specific outcome measures will be detailed in future subprojects.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Janne Vehreschild, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Ehren K, Hertenstein C, Kummerle T, Vehreschild JJ, Fischer J, Gillor D, Wyen C, Lehmann C, Cornely OA, Jung N, Gravemann S, Platten M, Wasmuth JC, Rockstroh JK, Boesecke C, Schwarze-Zander C, Fatkenheuer G. Causes of death in HIV-infected patients from the Cologne-Bonn cohort. Infection. 2014 Feb;42(1):135-40. doi: 10.1007/s15010-013-0535-7. Epub 2013 Oct 1. PMID 24081925
- [Derived] Trickey A, Ingle SM, Boyd A, Gill MJ, Grabar S, Jarrin I, Obel N, Touloumi G, Zangerle R, Rauch A, Rentsch CT, Satre DD, Silverberg MJ, Bonnet F, Guest J, Burkholder G, Crane H, Teira R, Berenguer J, Wyen C, Abgrall S, Hessamfar M, Reiss P, d'Arminio Monforte A, McGinnis KA, Sterne JAC, Wittkop L; Antiretroviral Therapy Cohort Collaboration. Contribution of alcohol use in HIV/hepatitis C virus co-infection to all-cause and cause-specific mortality: A collaboration of cohort studies. J Viral Hepat. 2023 Sep;30(9):775-786. doi: 10.1111/jvh.13863. Epub 2023 Jun 20. PMID 37338017
- [Derived] Trickey A, Sabin CA, Burkholder G, Crane H, d'Arminio Monforte A, Egger M, Gill MJ, Grabar S, Guest JL, Jarrin I, Lampe FC, Obel N, Reyes JM, Stephan C, Sterling TR, Teira R, Touloumi G, Wasmuth JC, Wit F, Wittkop L, Zangerle R, Silverberg MJ, Justice A, Sterne JAC. Life expectancy after 2015 of adults with HIV on long-term antiretroviral therapy in Europe and North America: a collaborative analysis of cohort studies. Lancet HIV. 2023 May;10(5):e295-e307. doi: 10.1016/S2352-3018(23)00028-0. Epub 2023 Mar 20. PMID 36958365
- [Derived] Mathe PJG, Usadel S, Rieg S, Kern WV, Muller MC. Long-term follow-up after introduction of a systematic sexually transmitted infection screening program for men having sex with men living with HIV in a primary care setting: uptake, STI incidence, and risk factors for infection and reinfection. Infection. 2023 Aug;51(4):897-907. doi: 10.1007/s15010-022-01946-0. Epub 2022 Nov 9. PMID 36352322
- [Derived] Stecher M, Chaillon A, Stephan C, Knops E, Kohmer N, Lehmann C, Eberle J, Bogner J, Spinner CD, Eis-Hubinger AM, Wasmuth JC, Schafer G, Behrens G, Mehta SR, Vehreschild JJ, Hoenigl M. Drug Resistance Spread in 6 Metropolitan Regions, Germany, 2001-20181. Emerg Infect Dis. 2020 Oct;26(10):2439-2443. doi: 10.3201/eid2610.191506. PMID 32946725
- [Derived] Stecher M, Hoenigl M, Eis-Hubinger AM, Lehmann C, Fatkenheuer G, Wasmuth JC, Knops E, Vehreschild JJ, Mehta S, Chaillon A. Hotspots of Transmission Driving the Local Human Immunodeficiency Virus Epidemic in the Cologne-Bonn Region, Germany. Clin Infect Dis. 2019 Apr 24;68(9):1539-1546. doi: 10.1093/cid/ciy744. PMID 30169606
- [Derived] Stecher M, Chaillon A, Eberle J, Behrens GMN, Eis-Hubinger AM, Lehmann C, Jablonka A, Bogner J, Fatkenheuer G, Spinner CD, Wasmuth JC, Kaiser R, Mehta SR, Vehreschild JJ, Hoenigl M. Molecular Epidemiology of the HIV Epidemic in Three German Metropolitan Regions - Cologne/Bonn, Munich and Hannover, 1999-2016. Sci Rep. 2018 May 1;8(1):6799. doi: 10.1038/s41598-018-25004-8. PMID 29717148
- See also: Related Info — http://www.dzif.de/en/research/hiv/